CLINICAL TRIAL: NCT00001540
Title: The Use of Bacteriophage Phi X174 to Assess the Immune Competence of HIV-Infected Patients In Vivo
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960058; 96-I-0058
Record Dates: First submitted 2000-04-01; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-02

CONDITIONS: HIV Infections
Keywords: Diagnostic; Immune Function; Immunization; Immunodeficiency; Quantitative
MeSH Terms: conditions — HIV Infections; Disease; Immunologic Deficiency Syndromes

SUMMARY:
The objective of this study is to evaluate the safety and utility of bacteriophage phi X174 immunization as a tool to assess the immune competence of HIV-infected patients at different stages of disease in vivo, and to assess the impact of viral load levels and therapy-induced changes in viral load levels on the response to immunization with the neo-antigen bacteriophage phi X174. Bacteriophage phi X174 immunization is a method that has been in use for more than 25 years to assess the immunity of patients with various types of primary and secondary immunodeficiencies, including 48 HIV-infected patients. This is a prospective open-label, controlled study which will enroll 39 HIV-infected patients and 13 healthy volunteers, male or female with 18 years of age and over. The HIV-infected patients will be divided into 3 groups according to their CD4 cell count: less than 200 cells/mm(3), between 200 and 500 cells/mm(3) and greater than 500 cells/mm(3). After screening and a two week pre-study evaluation, all eligible participants will receive a primary, secondary and tertiary immunization with 2 x 10(9) PFU/kg of bacteriophage phi X174 six weeks apart. Patients who present with detectable levels of viral load at entry will be offered a more effective antiviral drug regimen. Patients will have to be on a stable antiviral regimen for at least one month prior to receiving the primary immunization. Patients will return for visits 1, 2 and 4 weeks after each immunization for clinical and laboratory evaluations. The study endpoints are: safety (as measured by incidence of adverse events, CD4 cell count and HIV plasma RNA), kinetics of bacteriophage clearance following primary immunization, quantitation of bacteriophage phi X174 specific antibody titers following primary, secondary and tertiary immunizations and determination of qualitative and quantitative antibody isotype switching following secondary and tertiary immunizations.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and utility of bacteriophage phi X174 immunization as a tool to assess the immune competence of HIV-infected patients at different stages of disease in vivo, and to assess the impact of viral load levels and therapy-induced changes in viral load levels on the response to immunization with the neo-antigen bacteriophage phi X174. Bacteriophage phi X174 immunization is a method that has been in use for more than 25 years to assess the immunity of patients with various types of primary and secondary immunodeficiencies, including 48 HIV-infected patients. This is a prospective open-label, controlled study which will enroll 39 HIV-infected patients and 13 healthy volunteers, male or female with 18 years of age and over. The HIV-infected patients will be divided into 3 groups according to their CD4 cell count: less than 200 cells/mm(3), between 200 and 500 cells/mm(3) and greater than 500 cells/mm(3). After screening and a two week pre-study evaluation, all eligible participants will receive a primary, secondary and tertiary immunization with 2 x 10(9) PFU/kg of bacteriophage phi X174 six weeks apart. Patients who present with detectable levels of viral load at entry will be offered a more effective antiviral drug regimen. Patients will have to be on a stable antiviral regimen for at least one month prior to receiving the primary immunization. Patients will return for visits 1, 2 and 4 weeks after each immunization for clinical and laboratory evaluations. The study endpoints are: safety (as measured by incidence of adverse events, CD4 cell count and HIV plasma RNA), kinetics of bacteriophage clearance following primary immunization, quantitation of bacteriophage phi X174 specific antibody titers following primary, secondary and tertiary immunizations and determination of qualitative and quantitative antibody isotype switching following secondary and tertiary immunizations.

ELIGIBILITY:
Male or female; 18 years of age and over.

Women of child bearing potential must have a negative pregnancy test 2 weeks prior to immunization and must agree to use an active form of birth control during participation. Men should exercise appropriate contraceptive measures while participating on the study.

Ability and willingness to sign an informed consent.

Adequate venous access as assessed by the Principal or Associate Investigators.

Willingness to comply with the protocol requirements and visit schedule.

HIV-INFECTED PATIENTS:

HIV seropositivity on Elisa, confirmed with Western Blot.

No use or a stable use of an FDA-approved antiviral drug regimen for at least one month.

Life expectancy greater than 6 months.

NORMAL VOLUNTEERS:

Healthy (all clinical and laboratory tests should be in the normal range).

HIV seronegativity.

No signs and/or other laboratory evidence of immunodeficiency. These include a history of persistent or recurrent infections, infections with unusual organisms or autoimmunity.

No prior immunization with bacteriophage phi X 174.

No current active opportunistic infection.

No use of immune -based therapies or other experimental agents, corticosteroids (at doses greater than 25 mg/d of prednisone for more than 4 weeks) or any other immunosuppressive drugs within 6 months prior to enrollment.

No history of severe asthma defined by the need for intermittent or continuous corticosteroid therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52
Dates: Start 1996-04; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernstein LJ, Ochs HD, Wedgwood RJ, Rubinstein A. Defective humoral immunity in pediatric acquired immune deficiency syndrome. J Pediatr. 1985 Sep;107(3):352-7. doi: 10.1016/s0022-3476(85)80505-9. PMID 4032129
- [Background] Ochs HD, Junker AK, Collier AC, Virant FS, Handsfield HH, Wedgwood RJ. Abnormal antibody responses in patients with persistent generalized lymphadenopathy. J Clin Immunol. 1988 Jan;8(1):57-63. doi: 10.1007/BF00915157. PMID 2966810